CLINICAL TRIAL: NCT03773679
Title: The Effect of Daily Exercise Program on Bone Mineral Density and Cortisol Level in Preterm Infants With Very Low Birth Weight: A Randomized Controlled Trial
Brief Title: The Effect of Daily Exercise Program on Bone Mineral Density and Cortisol Level in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yağmur Sezer Efe, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016/282
Record Dates: First submitted 2018-12-03; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Osteopenia of Prematurity
Keywords: Preterm infants with very low birth weight (VLBW); bone mineral density; cortisol; exercise
MeSH Terms: conditions — Bone Diseases, Metabolic; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Daily exercise program involved "Range of Motion (ROM) exercises against extremity resistances" and "extension and flexion in upper and lower extremities." Exercises were implemented on wrists, elbows, shoulders, ankles, knees, and hip joints of the infants by the same researcher (YSE). The daily exercise program was repeated 5-8 times, 1 session/day (a similar time of the day), for 30 days. Each session continued for 7-10 minutes.
  Interventions: Procedure: Daily Exercise
- Control Group (No Intervention): The preterm infants in the control group did not receive the daily exercise program, only the standard clinical routine.

INTERVENTIONS:
Procedure: Daily Exercise — Daily Exercise Programme
  Arms: Exercise Group

SUMMARY:
ABSTRACT Objective: This randomized controlled double-blinded experimental study was carried out to determine the effects of daily exercise program on bone mineral density and cortisol level in preterm infants with very low birth weight matched for birth weight, gestation week, and gender.

Study design: The study was performed with preterm infants hospitalized in the neonatal intensive care unit of a tertiary hospital. Ethical committee approval, institutional permission, parental written consent were obtained. Daily exercise program was implemented in preterm infants in the exercise group for 30 days, once a day, and continuing for 7-10 minutes. Before and after the study the following were evaluated in preterm infants in the exercise and control group: anthropometric measurements, tibia speed of sound (SOS) for bone mineral density, serum biochemical parameters and cortisol levels.

DETAILED DESCRIPTION:
Objective: This randomized controlled double-blinded experimental study was carried out to determine the effects of daily exercise program on bone mineral density and cortisol level in preterm infants with very low birth weight matched for birth weight, gestation week, and gender.

Study design: The study was performed with preterm infants hospitalized in the neonatal intensive care unit of a tertiary hospital. Ethical committee approval, institutional permission, parental written consent were obtained. Daily exercise program was implemented in preterm infants in the exercise group for 30 days, once a day, and continuing for 7-10 minutes. Before and after the study the following were evaluated in preterm infants in the exercise and control group: anthropometric measurements, tibia speed of sound (SOS) for bone mineral density, serum biochemical parameters and cortisol levels.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria for the infants were as follows:

* postnatal age of 1-5 days,
* gestational age of 28-32 weeks,
* birth weight of 1,000-1,500 gr,
* no diagnosis of necrotizing enterocolitis (NEC), digestive system or chromosomal abnormalities, skin diseases, intrauterine growth retardation (IUGR), SGA, and large gestational age (LGA),
* no history of surgical intervention, and
* no medical treatment except for appropriate vitamin supplements and antibiotic treatments.

Exclusion Criteria:

-

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-04-15 (Actual); Primary Completion 2016-04-15 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Bone speed of sound values | Change from bone speed of sound values at 30 days
  To measure SOS values, the preterm infant was placed on his/her back and his/her right leg was placed to obtain an angle of 900. The middle of the medial malleolus and distal patella apex was found and then gel was poured between the skin and the probe. The probe was put parallel to the bone to contact the point determined to be in the middle of the tibia and was moved from inside the leg. Afterward, the probe was placed from outside the leg toward the inside. In this study, The SOS from tibia was measured.

SECONDARY OUTCOMES:
Serum Cortisol levels | Change from serum cortisol levels at 30 days
  serum biochemical parameters

CONTACTS AND LOCATIONS:
Overall Officials: Yagmur Sezer Efe, Principal Investigator — TC Erciyes University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sezer Efe Y, Erdem E, Gunes T. The Effect of Daily Exercise Program on Bone Mineral Density and Cortisol Level in Preterm Infants with Very Low Birth Weight: A Randomized Controlled Trial. J Pediatr Nurs. 2020 Mar-Apr;51:e6-e12. doi: 10.1016/j.pedn.2019.05.021. Epub 2019 Jul 6. PMID 31285069